CLINICAL TRIAL: NCT03590678
Title: Prospective Collection of Whole Blood Specimens in Pregnant Women
Brief Title: Collection of Whole Blood Specimens in Pregnant Women
Status: Completed | Type: Observational
Sponsor: Illumina, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RGH-015
Record Dates: First submitted 2017-05-04; First posted 2018-07-18 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Human blood specimens will be spun to plasma and stored at -80C freezers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Subject is scheduled for an invasive procedure and did not have NIPT testing in current pregnancy
- 2: Subject is scheduled for an invasive procedure and has a known positive or no-call result from a targeted NIPT in the current pregnancy

SUMMARY:
To prospectively collect whole blood specimens and clinical data from pregnant women scheduled for an invasive prenatal diagnostic procedure ("invasive procedure"). Specimens will be used for future testing with an investigational NIPT.

DETAILED DESCRIPTION:
This is a prospective multicenter study in which whole blood specimens will be collected from pregnant women scheduled for an invasive procedure.

After the standard-of-care invasive procedure is performed in accordance with the site's clinical procedures, invasive prenatal diagnostic procedure results will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older at enrollment,
* Has a viable pregnancy (with documented fetal heartbeat) of at least 10 weeks, 0 days gestation at the time of maternal specimen collection,
* Be scheduled for an invasive prenatal diagnostic procedure (either chorionic villus sampling [CVS], amniocentesis, or percutaneous umbilical cord blood sampling [cordocentesis]) for cytogenetic analysis of the fetus

Exclusion Criteria:

* Has a known maternal chromosomal anomaly,
* Had an invasive prenatal diagnostic procedure in the current pregnancy before maternal specimen collection
* Has a history of transplant or malignancy, or
* Had a transfusion of blood or blood components up to 8 weeks before maternal whole blood specimen collection
* Already participated in this study (enrolled previously).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with a viable pregnancy of at least 10 weeks, 0 days gestation who are scheduled for an invasive procedure performed per the standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Collect Whole Blood Specimens in Pregnant Women | 3 years
  To collect maternal whole blood specimens from approximately 5,150 women with corresponding cytogenetic results from invasive prenatal diagnostic procedures (performed per the standard of care) to achieve sample size goals

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Waldrep, MD, Principal Investigator — Medical City Dallas Hospital
Locations (16):
- United States (5):
  - Center for Fetal Medicine, Los Angeles, California
  - Maternal Fetal Medicine and Genetics, Riverside, California
  - Desert Perinatal Associates, Las Vegas, Nevada
  - Practice Research Organization, Dallas, Texas
  - Eastern Virgina Medical School, Dept Obstetrics and Gynecology, Maternal Fetal Medicine, Norfolk, Virginia
- Mater Misericordiae Limited, South Brisbane, Queensland, Australia
- Kuala Lumpur Hospital, Kuala Lumpur, Malaysia
- Poland (3):
  - Centrum Medyczne Angelius Provita, Katowice, Silesian Voivodeship
  - CENTRUM INNOWACYJNYCH TERAPII Sp. z, Piaseczno
  - FERTINA Sp. z o.o. SPÓŁKA KOMANDYTOWA, Warsaw
- Thailand (3):
  - Phramongkutklao Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Songklanagarind Hospital, Songkhla
- Ukraine (3):
  - "Institute of general practice - family medicine", Kyiv
  - LLC "Reproductive Genetics Clinic "Victoria", Kyiv
  - Medical Center "Pulse", Small Private Business, Vinnytsia

IPD SHARING:
Plan to Share IPD: No